CLINICAL TRIAL: NCT02202460
Title: The Potential Biomark of Serious Psychosis: Including the Variation of Brain MRI, BDNF and Oxidative Stress-related Immunological Factors in Different Phases.
Brief Title: The Potential Biomark of Serious Psychosis:a Prospective,Case-controled Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Renrong Wu, Professor, Central South University
Other Study IDs: rrw2014; IFMISMD (Registry Identifier: IFMISMD)
Record Dates: First submitted 2014-06-12; First posted 2014-07-29 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Other Immunological States or Disorders
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Patients suffer from Serious Psychosis may have variation in immunological factors,BDNF and MRI.

DETAILED DESCRIPTION:
Patients suffer from Schizophrenia and Mood Disorders may have variation in immunological factors(TNF-α,IL-2,IL-6,IL-10,etc),BDNF and Brain MRI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with Schizophrenia , Bipolar Disorder or Major Depression by DSM-5

Exclusion Criteria:

* Unstable physical conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Schizophrenia , Bipolar Disorder , Major Depression
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Oxidative Stress-related Immunological Factors | 18 month
  Blood test will be conducted every 3 month to assess the concentration of oxidative stress-related immunological factors including TNFα,TGFβ， MCP-1，IL-1α，IL-2，IL-6，IL-10，IL-12.

SECONDARY OUTCOMES:
BDNF | 18 month
  Collecting participants' blood every 3 month to assess the concentration of brain derived neurotrophic factor.

OTHER OUTCOMES:
Brain MRI | 18 month
  Brain MRI will be examined every 6 month or when onset syptoms are dramatically changed.

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Institute of 2nd Xiangya Hospital,CSU, Changsha, Hunan, China